CLINICAL TRIAL: NCT00241579
Title: Analgesic Efficacy of Smoked Cannabis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Medicinal Cannabis Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C00-SD-107; 021422
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2006-06

CONDITIONS: Pain; Hyperalgesia
Keywords: Pain; Cannabis; Analgesic
MeSH Terms: conditions — Pain; Hyperalgesia; Marijuana Abuse

INTERVENTIONS:
Drug: Smoked Cannabis

SUMMARY:
The purpose of this study is to determine whether or not inhaled marijuana displays any pain-relieving properties on experimentally-induced pain.

DETAILED DESCRIPTION:
It is important to evaluate the effects of the cannabinoids on facilitated pain as conditions of hyperalgesia more closely approximates the clinical situation. There are limited clinical studies on the effect of the cannabinoids on facilitated pain states. Noyes et al evaluated the analgesic effects of Delta-9-THC in 34 cancer patients with pain. They concluded that 20mg of oral Delta-9-THC was similar to 120mg of codeine (Noyes et al, 1975). Jain et al concluded that 1.5-3mg of intramuscular Levonantradol resulted in significant pain relief as compared to placebo in 56 patients with acute postoperative pain (Jain et al, 1981).

Comparison(s): Three different doses of smoked cannabis will be compared to placebo for the reduction of experimentally induced pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Male or Female
* Subject smoked cannabis within the last six months

Exclusion Criteria:

* Active opportunistic infections or opportunistic malignancies requiring acute treatment
* Active substance abuse (alcohol or injection drug)
* Pulmonary complications (e.g., tuberculosis, asthma)
* Current use of cannabis (e.g., within 30 days of randomization)
* Pregnancy as ascertained by a self-report and a mandatory commercial pregnancy test before any cannabis or placebo consumption condition
* Personal or familial history of psychiatric disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2002-02; Study Completion 2004-01

PRIMARY OUTCOMES:
Score on a Visual Analog Scale (VAS) of pain severity
McGill Pain Questionnaire (MPQ) Short Form
Neurosensory testing of: 1) warm and cold sensation, 2) warm and cold pain, 3) touch, and 4) mechanical pain. Testing administered using a Thermal Sensory Analyzer, von Frey hair filaments, and a pinch algometer, respectively.

SECONDARY OUTCOMES:
Trail Making Test (TMT) as a measure of psychomotor speed.
Paced Auditory Serial Attention Test (PASAT) as a measure of speed of information processing.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wallace, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Medical Center, San Diego, California, United States

REFERENCES:
- See also: Center for Medicinal Cannabis Research — http://cmcr.ucsd.edu